CLINICAL TRIAL: NCT02252146
Title: Phase I/II Open-label, Multiple-dose, Dose-escalation Study to Evaluate the Safety and Tolerability of IMO-8400 in Patients With Relapsed or Refractory Diffuse Large B-Cell Lymphoma and Presence of the MyD88 L265P Mutation
Brief Title: Dose Escalation Study in Patients With Relapsed or Refractory DLBCL and MyD88 L265P Mutation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Idera Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8400-402
Record Dates: First submitted 2014-08-08; First posted 2014-09-30 (Estimated); Results first posted 2017-11-14 (Actual); Last update posted 2017-12-12 (Actual); Status verified 2017-11

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: DLBCL; MYD88 L265P; Lymphoma; Diffuse Large B Cell Lymphoma; Idera; IMO 8400
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma | interventions — bazlitoran

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IMO-8400 (Experimental): IMO-8400 0.3 mg/kg twice weekly, 0.6 mg/kg twice weekly, or 1.2 mg/kg twice weekly
  Interventions: Drug: IMO-8400

INTERVENTIONS:
Drug: IMO-8400 — MO-8400 given subcutaneously twice weekly

SUMMARY:
Recent reports have identified a specific oncogenic mutation L265P of the MYD88 gene in approximately 30% of the patients with the activated B-cell (ABC) type of Diffuse Large B Cell Lymphoma (DLBCL). MYD88 is an initial adapter linker protein in the signaling pathway of the Toll Like Receptors (TLRs), including the endosomal TLRs 7, 8, and 9, for which the ligands are nucleic acids. IMO-8400 is an oligonucleotide specifically designed to inhibit ligand activation of TLRs 7,8, and 9. Recent studies indicate that in the presence of L265P mutation ligand activation of those TLRs results in markedly increased signaling with subsequent increased cell activation, cell survival, and cell proliferation. The scientific rationale for assessing the use of IMO-8400 to treat patients with DLBCL and the L265P mutation is based on laboratory observations that IMO-8400 inhibits ligand-based activation of cells with the mutation and decreases the survival and proliferation of the cell populations responsible for the propagation of the disease.

DETAILED DESCRIPTION:
Eligible subjects will be enrolled and assigned to one of five dose cohorts. Treatment will be administered by subcutaneous injection until progression or intolerable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of Diffuse Large B Cell Lymphoma (DLBCL) of non-GCB subtype, established according to the World Health Organization (WHO) criteria that has been tested for the MyD88 L265P mutation.
* In addition to the above, key inclusion and exclusion criteria are listed below.

  1. Be at least 18 years of age
  2. Agree to use contraception

Exclusion Criteria:

1. Is nursing or pregnant
2. DLBCL of GCB subtype
3. Has BMI > 34.9 kg/m2
4. Has a positive test for human immunodeficiency virus (HIV-1 or -2) hepatitis C virus (HCV) or hepatitis B surface antigen (HBsAg)
5. Receiving chronic systemic corticosteroid therapy > 20 mg of prednisone daily
6. Being treated with other anti-cancer therapies (approved or investigational)
7. Has an active infection requiring systemic antibiotics
8. Has had surgery requiring general anesthesia within 4 weeks of starting the study
9. Has heart failure of Class III or IV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-06; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Cornfeld, MD, MPH, Study Director — Idera Pharmaceuticals, Inc.
Locations (12):
- United States (12):
  - UCLA Medical Center, Los Angeles, California
  - Emory University, Atlanta, Georgia
  - Cancer Care Specialists of Illinois, Decatur, Illinois
  - Horizon Bio Advance, Lafayette, Indiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Columbia University Medical Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Vanderbilt Ingram Cancer Center, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- IMO-8400: IMO-8400 0.3 mg/kg twice weekly, 0.6 mg/kg twice weekly, or 1.2 mg/kg twice weekly
  IMO-8400: IMO-8400 given subcutaneously twice weekly
Period: Overall Study
Arm/Group | IMO-8400
Started | 6
Completed | 0
Not Completed | 6
Not completed — Lack of Efficacy | 4
Not completed — Entered hospice care | 1
Not completed — Inability to travel to study site | 1

BASELINE CHARACTERISTICS:
Population: Safety population
Arm/Group | IMO-8400
Number analyzed (Participants) | 6
Age, Continuous [Median (Full Range); unit: years] | 67 [61 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events, Injection Site Reactions, and Concomitant Medications
Description: Frequency of adverse events, injection site reactions, and concomitant medications observed
Time Frame: Up to 2 years from first patient visit
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | IMO-8400
Number analyzed (Participants) | 6
Participants
  Subjects with TEAEs | 4
  Subjects with ISRs | 1
  Subjects with Concomitant Medications | 3

ADVERSE EVENTS:
Time Frame: Up to 2 years after start of study treatment
Arm/Group | IMO-8400
All-Cause Mortality (participants affected / at risk) | 1/6
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IMO-8400 (N=6)
Abdominal pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Disease progression (General disorders) | 1
Pyrexia (General disorders) | 1
Sepsis (Infections and infestations) | 1
Radiation necrosis (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IMO-8400 (N=6)
Anemia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Lacrimation increase (Eye disorders) | 2
Dry eye (Eye disorders) | 1
Eye discharge (Eye disorders) | 1
Eye pain (Eye disorders) | 1
Ocular hyperaemia (Eye disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 1
Disease progression (General disorders) | 1
Injection site reaction (General disorders) | 1
Pyrexia (General disorders) | 1
Oral herpes (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Radiation necrosis (Injury, poisoning and procedural complications) | 1
Neutrophil count decreased (Investigations) | 1
Weight decreased (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Investigations) | 1
Hyponatraemia (Investigations) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Lethargy (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Hypotension (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-01-29): https://cdn.clinicaltrials.gov/large-docs/46/NCT02252146/Prot_000.pdf
  • Statistical Analysis Plan (2016-11-11): https://cdn.clinicaltrials.gov/large-docs/46/NCT02252146/SAP_001.pdf